CLINICAL TRIAL: NCT07301853
Title: Longitudinal Follow-up and Health-Related Outcomes in Liver Transplant Recipients and Living Donors
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Mukogawa Women's University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-0793
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Living Donor Liver Transplantation Recipients; Deceased Donor Liver Transplantation Recipients; Living Liver Donor
Keywords: liver transplantation; living donors; transplant recipients; follow-up studies
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recipients: A patient who received a new, healthy liver (or part of one from a living donor) to replace their own diseased liver
  Interventions: Procedure: liver transplantation
- living donors: A healthy person who donated a portion of their healthy liver to someone with liver failure.
  Interventions: Procedure: Living Donor Hepatectomy

INTERVENTIONS:
Procedure: liver transplantation — Patients undergo standard liver transplantation according to clinical protocols. Postoperative management and follow-up are conducted per routine standard of care. Clinical data, including survival, adverse events, and quality of life (assessed by questionnaires/scales), are collected observationally at regular follow-up intervals.
  Groups: recipients
Procedure: Living Donor Hepatectomy — Living donors undergo standard hepatectomy procedures. Postoperative recovery and long-term health outcomes are monitored through routine follow-up visits and assessments.
  Groups: living donors

SUMMARY:
This prospective cohort study aims to identify risk factors for postoperative adverse events in liver transplant recipients and living donors. By collecting comprehensive clinical data and conducting systematic long-term follow-up, the researchers intend to establish a specialized, standardized, and individualized follow-up management system. The ultimate goal is to optimize intervention strategies and improve patient prognosis and quality of life for both recipients and donors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing liver transplantation or living donor hepatectomy at the study center (living donor should be approved by the hospital ethics committee for living organ donation);
2. Age 18 years or older;
3. Willing to participate in the long-term follow-up management program;
4. Signed informed consent form;

Exclusion Criteria:

1. Patients undergoing combined organ transplantation
2. Patients with severe mental illness or cognitive impairment who are unable to cooperate with follow-up assessments.
3. Donors whose surgery is aborted intraoperatively for any reason.
4. Unable or unwilling to comply with the long-term follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises all consecutive patients with end-stage liver disease or acute liver failure scheduled for liver transplantation (recipients) and healthy individuals undergoing living donor hepatectomy (donors) at the Department of Liver Surgery of the study center. Participants are selected from the clinical practice setting of the study center.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2045-12-31 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term Incidence of Postoperative Adverse Events | From date of surgery up to 20 years
  Evaluation of the cumulative incidence of postoperative complications

SECONDARY OUTCOMES:
Overall Survival | Up to 20 years
Graft Survival Rate | Up to 20 years
Patient-Reported Outcome questionnaire | Baseline and annually up to 20 years
  Assessment of multiple dimensions of patient health status, including physical functioning, mental health, social well-being, symptoms burden (e.g., pain, fatigue), and medication adherence. These domains will be evaluated using a battery of standard validated instruments

CONTACTS AND LOCATIONS:
Overall Officials: Wen Fang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China